CLINICAL TRIAL: NCT02185586
Title: A Prospective Randomized Controlled Trial of Traditional Three-port Laparoscopic Cholecystectomy Versus Lower Abdominal Three-port Laparoscopic Cholecystectomy
Brief Title: A Prospective Randomized Controlled Trial of Lower Abdominal Three-port Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Li Xu, Department of hepatobiliary surgery, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-21; 2014-21 (Other Grant/Funding Number: Ethic committee of China-Japan Friendship Hospital)
Record Dates: First submitted 2014-07-06; First posted 2014-07-09 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Gallbladder Stone; Gallbladder Polyp
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LALC (Experimental): lower abdominal laparoscopic cholecystectomy
  Interventions: Procedure: laparoscopic cholecystectomy
- SLC (Experimental): single laparoscopic cholecystectomy
  Interventions: Procedure: laparoscopic cholecystectomy
- UALC (Placebo Comparator): upper abdominal laparoscopic cholecystectomy
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy
  Other Names: lower abdominal three-port laparoscopic cholecystectomy; single port laparoscopic cholecystectomy; upper abdominal three-port laparoscopic cholecystectomy

SUMMARY:
We have designed a new method which could be used in laparoscopic cholecy- stectomy.Account to this new method, the three incisions are all located on the lower abdominal, theoretically it could get more beautiful outlook and less stress response than traditional laparoscopic cholecystectomy(two of the three incisions located on upper abdomen) or single port laparoscopic cholecystectomy(one large incision located on umbilicus).

We plan to conduct a randomized controlled trial to compare those there methods of laparoscopic cholecystectomy, in order to find out if there will be some advantages of this new method,such as in lowering the stress response,reducing impact on respiration, relieving post-operation pain and improving appearance.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 70 years old
* benign diseases of gallbladder
* selective cholecystectomy
* Capable to read and write

Exclusion Criteria:

* accept upper abdominal operation before
* acute cholecystitis
* with serious heart or pulmonary diseases
* with diseases of immune system
* Pregnant women
* can not understand the research purposes
* relatives of researchers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Systematic inflammatory response caused by the surgical trauma | one day before the operation,8 hours after the operation,one day after the operation
  Blood IL-6,TNF-α,and CRP levels determined by ELISA at different time-points,

SECONDARY OUTCOMES:
Cosmesis and body image score | 1 and 3 months after the operation
pulmonary function | one day before the operation, one day after the operation
Post-operation pain score (visual analog scale, VAS) | 12 and 24 hours after the operation
36-item health survey | 3 months after the operation

OTHER OUTCOMES:
perioperative indexes | perioperative period
  operative duration,intra-operative blood loss, indication for additional trocar placement or conversion to open surgery, postoperative complications and duration of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, MD, Principal Investigator — China-Japan Friednship Hospital
Locations (1):
- Department of hepatobiliary surgery,China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided